CLINICAL TRIAL: NCT01178398
Title: A Qualitative Study of Fish Consumption During Pregnancy
Brief Title: Understanding Fish Consumption Habits During Pregnancy
Status: Completed | Type: Observational
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Emily Oken, Professor, Harvard Pilgrim Health Care
Other Study IDs: 0613; P30ES000002 (NIH)
Record Dates: First submitted 2010-08-03; First posted 2010-08-10 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2010-08

CONDITIONS: Nutrition
Keywords: fish; pregnancy; nutrition; mercury; focus group; omega-3 fatty acid; docosahexaenoic acid (DHA)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Many pregnant women in the US do not consume enough docosahexaenoic acid (DHA), an essential nutrient found in fish. Apparently conflicting findings that fish consumption is beneficial for the developing fetus, yet potentially toxic because of mercury contamination, have created uncertainty about the appropriate fish consumption advice to provide pregnant women. The investigators objective was to determine knowledge, behaviors, and received advice regarding fish consumption among pregnant women who are infrequent consumers of fish.

DETAILED DESCRIPTION:
Fish is a healthful food that is the primary dietary source of elongated n-3 polyunsaturated fatty acids (PUFA), nutrients essential for optimal neurodevelopment. Most pregnant women in the US do not consume adequate n-3 PUFA. However, fish also may be contaminated with methylmercury, and approximately 10% of women of childbearing age in the US have mercury levels higher than recommended. Because the same food contains both essential nutrients and harmful contaminants, substantial confusion reigns about the best course of action for pregnant women. Additionally, it is not clear what fish consumption advice would be most effective in changing women's fish consumption habits. The goal of this pilot study is to perform formative work to allow us to develop and refine an intervention to promote consumption of fish low in mercury and high in n-3 PUFA among pregnant women. This project, together with a pilot RCT already funded, will serve as preliminary data to support a larger RCT to evaluate the effects of the intervention on pregnancy outcomes and postpartum maternal and infant health.

Specific Aims Aim 1. Among pregnant women, identify: 1) knowledge of the potential risks and benefits associated with fish consumption during pregnancy; 2) awareness of current recommendations for fish consumption by pregnant women; 3) the sources of information from which they are learning about the health effects associated with fish intake; and 4) facilitators and barriers to fish consumption, such as cost, availability, taste, and habits. To achieve this aim, we will conduct focus groups with pregnant women in the Boston area who are infrequent consumers of fish (defined as <= 2 monthly fish servings).

Aim 2. Develop materials for a planned intervention to increase consumption of fish high in n-3 polyunsaturated fatty acids and low in methylmercury among pregnant women who are infrequent consumers of fish at baseline. We will use results from Aim 1 to inform the development of these materials.

ELIGIBILITY:
Inclusion Criteria:

* currently pregnant
* age at least 18 years

Exclusion Criteria:

* unable to speak or understand English
* consuming 2 or more weekly fish servings
* unable to eat fish (e.g. allergy, dietary restriction)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women aged 18+ who are currently pregnant and who consume <2 weekly fish servings
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Oken, MD, MPH, Principal Investigator — Harvard Pilgrim Health Care Institute
Locations (1):
- Harvard Pilgrim Health Care Institute, Boston, Massachusetts, United States